CLINICAL TRIAL: NCT02694887
Title: Agreement Between Capillary and Venous Lactate in Emergency Department Patients
Brief Title: Capillary and Venous Lactate in Emergency Department Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Colin Graham, Professor, Chinese University of Hong Kong
Other Study IDs: CRE- 2015.624
Record Dates: First submitted 2016-02-12; First posted 2016-03-01 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Triage Category 3 (Urgent)
Keywords: Capillary blood; Venous blood; Lactate; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the present project is to study the accuracy of capillary blood level measured by handheld lactate analyzers when compared with the reference methods e.g.venepuncture blood gas analyzer sample.

DETAILED DESCRIPTION:
Background:

Increase in lactate levels (hyperlactataemia) is common in critically ill patients and it is a sensitive marker in early identification of patients who are critically ill. Blood lactate is also a predictor of clinical outcomes. High level of lactate is associated with high mortality as well as increased morbidity. Capillary blood sample is easy to collect, less painful, and its measurement using handheld device which may allow more rapid determination of test results in ED. This rapid lactate measurement could aid early recognition of patients at high risk of mortality and morbidity. However, the accuracy of this rapid capillary lactate measurement using handheld devices has not been well studied in ED patients.

Objective:

To study the accuracy of capillary blood level measured by handheld lactate analyzers when compared with the reference methods e.g.venepuncture blood gas analyzer sample.

Study design:

This is a prospective observational study of patients presenting to ED of Prince of Wales Hospital (PWH). Patients aged 18 or above who are triage category 3 presenting to ED will be recruited. Capillary and venous blood samples will be collected. Venous lactate levels will be measured by blood gas analyzer (Siemens Automatic QC RAPID Systems RAPID Point@500) and two hand-held lactate analyzers (StatStrip Xpress Lactate Meter and Lactate Scout + ). Venous lactate levels measured by blood gas analyzer will be served as "reference method". Capillary lactate levels will be analyzed by handheld lactate analyzer. We are aimed to recruited 240 patients.

Outcomes:

The primary outcome is the accuracy of capillary blood level measured by handheld lactate analyzers when compared with the reference methods e.g. venepuncture blood gas analyzer sample. The secondary outcomes are: (1) compare the difference in values of venous lactate using blood gas analyzer and hand-held lactate analyzers, (2) compare values of capillary and venous lactate using hand-held lactate analyzers, (3) compare the reporting times of handheld and blood gas analyzer, and (4) Compare values of capillary lactate using between the two hand-held lactate analyzers.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above who are triage category 3 in emergency department
* Presenting to emergency department between 9am and 4pm, Monday to Friday

Exclusion Criteria:

* Aged below 18 years
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or above who are triage category 3 presenting to Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02-08 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
The accuracy of capillary blood level measured by handheld lactate analyzer when compared with the reference methods e.g.venepuncture blood gas analyzer sample. | 30 minutes after recruitment

SECONDARY OUTCOMES:
Value of venous lactate measured using blood gas analyzer and handheld lactate analyzers | 30 minutes after recruitment
Value of venous lactate and capillary lactate measured using handheld lactate analyzers | 30 minutes after recruitment
Reporting time of venous lactate level measured using blood gas analyzer and reporting time of capillary lactate using hand-held lactate analyzers | 30 minutes after recruitment
Value of capillary lactate measured using two hand-held lactate analyzers | 30 minutes after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Graham, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Graham CA, Leung LY, Lo RS, Lee KH, Yeung CY, Chan SY, Cattermole GN, Hung KK. Agreement between capillary and venous lactate in emergency department patients: prospective observational study. BMJ Open. 2019 Apr 3;9(4):e026109. doi: 10.1136/bmjopen-2018-026109. PMID 30948594